CLINICAL TRIAL: NCT02888418
Title: Random, Double Blind, Placebo Controlled Phase I Clinical Trials to Estimate the Safety and Preliminary Immunogenicity of Tetravalent Recombinant Human Papilloma Virus Vaccine (6,11,16,18 Type)(Hansenula Polymorpha) in Women of 9 to 30 Years Old and Men of 9 to 17 Years Old
Brief Title: Safety and Immunogenicity Study of Human Papilloma Virus Vaccine in Women Aged 9 to 30 and Men Aged 9 to 17
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: cycdc2016-4
Record Dates: First submitted 2016-08-11; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Cervical Cancer
Keywords: vaccine; safety; immunogenicity
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- One dose of HPV vaccine in women aged 18 to 30 (Experimental): One dose of Tetravalent recombinant human papilloma virus vaccine (6,11,16,18 type) (Hansenula polymorpha) in women aged 18 to 30.
  Interventions: Biological: Tetravalent recombinant human papilloma virus vaccine (6,11,16,18 type) (Hansenula polymorpha)
- Placebo in women aged 18 to 30 (Placebo Comparator): Placebo in women aged 18 to 30.
  Interventions: Biological: placebo
- One dose of HPV vaccine in women aged 9 to 17 (Experimental): One dose of Tetravalent recombinant human papilloma virus vaccine (6,11,16,18 type) (Hansenula polymorpha) in women aged 9 to 17.
  Interventions: Biological: Tetravalent recombinant human papilloma virus vaccine (6,11,16,18 type) (Hansenula polymorpha)
- Placebo in women aged 9 to 17 (Placebo Comparator): Placebo in women aged 9 to 17.
  Interventions: Biological: placebo
- One dose of HPV vaccine in men aged 9 to 17 (Experimental): One dose of Tetravalent recombinant human papilloma virus vaccine (6,11,16,18 type) (Hansenula polymorpha) in men aged 9 to 17.
  Interventions: Biological: Tetravalent recombinant human papilloma virus vaccine (6,11,16,18 type) (Hansenula polymorpha)
- Placebo in men aged 9 to 17 (Placebo Comparator): Placebo in men aged 9 to 17.
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Tetravalent recombinant human papilloma virus vaccine (6,11,16,18 type) (Hansenula polymorpha) — Injection vaccine produced by Beijing institute of biological products co., LTD, containing HPV antigen protein, 120μg/0.5ml/bottle
  Arms: One dose of HPV vaccine in men aged 9 to 17; One dose of HPV vaccine in women aged 18 to 30; One dose of HPV vaccine in women aged 9 to 17
Biological: placebo
  Arms: Placebo in men aged 9 to 17; Placebo in women aged 18 to 30; Placebo in women aged 9 to 17

SUMMARY:
This study evaluates the safety of Tetravalent recombinant human papilloma virus vaccine (6,11,16,18 type) (Hansenula polymorpha) in women of 9 to 30 years old and men of 9 to 17 years old and preliminarily explore the immunogenicity.

135 people are enrolled in total, including 45 women of 18 to 30 years old and 90 people of 9 to 17 years old. Among the first group, 30 women will be inoculated studied vaccine and 15 women will be inoculated placebo. Among the second group, there are 45 women and 45 men, 30 women and 30 men in vaccine group and 15 women and 15 men in placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Requirements of age: males of 9 to 17 years old, females of 9 to 30 years old.
* Willing to provide the statutory certificate of identity.
* For subjects of 18 to 30 years old, they should be able to understand the clinical trials and agreed to sign the informed consent; for subjects of 9 to 17 years old, their guardian should be able to understand the clinical trial, and sign informed consent together with subjects.
* Female subjects have no pregnancy and birth plans in the 7 months after being enrolled, and agree to take effective contraception during this period.

Exclusion Criteria:

* People with history of cervical cancer or HPV infection related diseases such as condyloma
* People with a history of severe allergic reactions requiring medical intervention (such as garget, difficult breathing, hypotension or shock)
* People with a history of serious side effects after vaccination or severe allergic reaction to food or drugs
* People with epilepsy or a history of mental illness
* People in immune deficiency or diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases, people with immunosuppressive therapy in the past six months.
* People with serious liver or kidney disease, cardiovascular disease, severe hypertension, diabetes, cancer, all kinds of infectious disease and acute disease or in acute attack period of chronic diseases
* Asplenia, functional asplenia, and any situation leading to asplenia or splenectomize.
* People diagnosed by doctors with coagulation dysfunction (such as the lack of clotting factors, disorders of blood coagulation and blood platelet disorders), apparent bruises or blood coagulation disorders;
* People given whole blood, plasma or immunoglobulin therapy within 3 months before vaccination.
* People get any vaccine within 14 days before the trial.
* People with fever before vaccination, axillary temperature higher than 37.0 ℃.
* Females in suckling period, pregnancy (pregnancy test positive) or prepared to be pregnant.
* People with abnormal laboratory index. (slight abnormity is except if judged with no clinical significance by doctors.)
* People has gotten HPV vaccine before; people has used or plans to use other vaccine or unregistered products (drugs or vaccines) within 30 days before the first dose; people plans to participate in other clinical trials within 6 months after this clinical trial.
* According to judgement of researchers, the subjects have any other factors that are not appropriate for this clinical trials.

The exclusion criteria for the second and third dose：

* Urine pregnancy test are positive before vaccination.
* Receiving blood products or other studied drugs after enrollment.
* Suffering from serious illness or with serious adverse events that require continuous treatment.
* Situations need to be excepted according to the judgement of researchers or the confirmation of Ethics Committee.
* Newly occurred or discovered people that does not meet exclusion criteria of first dose after the first vaccination.

Delayed immunization:

* Acute infectious disease, temperature being over 37.0 ℃or acute attack of chronic disease before inoculation.
* Physical examination is abnormal on the day of vaccination.
* Researchers think that the subjects belong to other temporary contraindications of vaccination.

Withdrawal criteria:

* Any situation in exclusion criteria after enrollment.
* People who suffers from diseases that need to be treated by immune inhibitors should be dropped out, in case of the harm of diseases that need to be treated by immune inhibitors.
* Serious adverse events: events that need or prolong hospitalization, disability, threatening lives or death. Researchers decide whether to quit the trial.
* Against the plan and deviation from the plan:

  1. against the plan events

     * no appropriate informed consent for the subjects;
     * the subjects get into the research while do not meet the inclusion criteria or meet the exclusion criteria.
     * subjects use the vaccines that are not preserved as requested.
     * serious adverse event (SAE) does not be reported or timely reported.
     * subjects proactively use forbidden drugs (anti-allergic drug, antipyretic and analgesic, accepting systemic corticosteroids more than 2 mg/kg/day by intramuscular injection, oral or intravenous administration, continuing more than 14 days, or other immune inhibitors).
  2. deviation from the plan

     * exceeding the Window of supervision.
     * the blood sample of subjects does not be collected or sample quantity is not enough to finish the test.
     * no enough interval with other vaccines.

Ages: 9 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 135 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Rate of Adverse reactions of Human Papilloma Virus Vaccine in Women Aged 9 to 30 and Men Aged 9 to 17 | 30 days
  Adverse reactions associated with vaccine will be observed in subjects after vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy.

SECONDARY OUTCOMES:
Evaluate the seroconversion rate of HPV antibodies in serum after vaccination. | 30 days
  The seroconversion rate will be evaluated at 30 days after vaccination.